CLINICAL TRIAL: NCT04420377
Title: The Chronic Effects of L-Carnitine Tartrate Supplementation on Recovery
Brief Title: The Chronic Effects of Carnitine on Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Applied Science & Performance Institute (Industry)
Collaborators: Lonza Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0220
Record Dates: First submitted 2020-05-20; First posted 2020-06-09 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Muscle Soreness; Muscle Damage; Resistance Training; Oxidative Stress; Muscle Strength
Keywords: Ergogenic Aid; Muscle Recovery; Resistance Training
MeSH Terms: conditions — Myalgia | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: Double-blind, parallel, randomized, placebo-controlled trial.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Group (Placebo Comparator): Participants will engage in a 5-week, whole-body, resistance training program 2 days per week will consuming a visually identical placebo (25mg hydroxypropyl methylcellulose) 30 minutes prior to exercise on training days or with the first meal of the day on non-training days. For week 5 of the study, participants will come in for 1 intense exercise training day.
  Interventions: Other: Resistance Training
- Experimental Group (Experimental): Participants will engage in a 5-week, whole-body, resistance training program 2 days per week will consuming a treatment condition (Carnipure™) 30 minutes prior to exercise on training days or with the first meal of the day on non-training days. For week 5 of the study, participants will come in for 1 intense exercise training day.
  Interventions: Dietary Supplement: Carnipure; Other: Resistance Training

INTERVENTIONS:
Dietary Supplement: Carnipure — Supplement contains L-carnitine tartrate.
  Arms: Experimental Group
Other: Resistance Training — 5 weeks of whole-body resistance training, performed 2 times per week.

SUMMARY:
This study investigated the effects of CarnipureTM, a high-quality L-carnitine ingredient, on long term (5 weeks) recovery, muscle damage, and SOD status in a population of males and females while training two days per week. The primary outcomes defining recovery were changes in serum creatine kinase levels and perceptual changes in recovery. Supporting variables included an assessment of strength and power as a functional indicator of recovery. This study would be the first to examine the effects of CarnipureTM on long-term recovery. Our primary hypothesis was that L-carnitine supplementation would reduce muscle damage and improve perceptual measures of recovery. Our secondary hypotheses were that L-carnitine supplementation would better sustain strength and power and elevate SOD status.

DETAILED DESCRIPTION:
This study investigated the effects of CarnipureTM, a high-quality L-carnitine ingredient, on long term (5 weeks) recovery, muscle damage, and SOD status in a population of males and females while training two days per week. The primary outcomes defining recovery were changes in serum creatine kinase levels and perceptual changes in recovery. Supporting variables included an assessment of strength and power as a functional indicator of recovery. This study would be the first to examine the effects of CarnipureTM on long-term recovery. Our primary hypothesis was that L-carnitine supplementation would reduce muscle damage and improve perceptual measures of recovery. Our secondary hypotheses were that L-carnitine supplementation would better sustain strength and power and elevate SOD status.

In totality, the study will last 5-weeks, consisting of supplementation with maintenance exercise performed 2 days per week, at home. Week 5 will consist of a pre-training assessment, an intense lower-body strength endurance training day, and subsequent testing 48-hour testing (Post-Week 5). The baseline testing (will be performed on approximately 10 subjects per day over the course of 4 days) and will consist of the following measures:

* DEXA (Dual Energy X-ray Absorptiometry) Body Composition Analysis
* Blood Draw
* Salivary Measures
* Isometric Mid Thigh Pull
* Force Plate Mechanography
* Visual Analog Scales

For the first 4 weeks of training, participants will be asked to workout 2 days per week at home.

On Monday of week five, 20 subjects will be assessed on the following measures:

* DXA
* Blood Draw
* Salivary Measures
* Isometric Mid Thigh Pull
* Force Plate Mechanography
* Visual Analog Scales

On Tuesday of week 5, the 20 subjects that tested on Monday, will go through an intense lower body, strength endurance protocol, and the leftover 20 subjects will go through the following assessments:

* DXA
* Blood Draw
* Salivary Measures
* Isometric Mid Thigh Pull
* Force Plate Mechanography
* Visual Analog Scales
* Before and After the workout - Finger Prick Blood Sample

On Wednesday of week 5, the 20 subjects that tested Monday, will have a day to rest. The 20 subjects that tested Tuesday, will go through an intense lower body strength endurance protocol.

* Before and After the workout - Finger Prick Blood Sample (for blood lactate)

On Thursday of week 5, the 20 subjects that tested Tuesday will have the day off, while the 20 subjects that tested Monday will be assessed on the following measures:

* Blood Draw
* Salivary Measures
* Isometric Mid Thigh Pull
* Force Plate Mechanography
* Visual Analog Scales

On Friday of week 5, the 20 subjects that tested Tuesday will be assessed on the following measures:

* Blood Draw
* Salivary Measures
* Isometric Mid Thigh Pull
* Force Plate Mechanography
* Visual Analog Scales

Participation will be sought from 80 male and female subjects ranging from 21 to 65 years old who are active (i.e. 30 minutes per week of moderate activity classified as greater than 50 % of their heart rate (HR) max 3 days • week-1). Two cohorts of 40 subjects will be examined in the study.

The supplement will be administered as a dose of 2g of Carnipure (L-carnitine), per day for the duration of the study. Placebo and treatment conditions will be administered in visually identical capsules. Statistical analysis will be carried out on the entire study population and on the female study population independently.

ELIGIBILITY:
Inclusion Criteria:

- Participation in at least 30 minutes of moderate activity exercise 3 times per week

Exclusion Criteria:

* Body-mass index (BMI) of ≥ 30 kg/m²;
* Cardiovascular, metabolic, endocrine, or thyroid disease
* Smoking tobacco
* Drinking alcohol (>7 or >14 drinks per week for women and men, respectively)
* Pregnancy
* Hypertension
* Hyperlipidemia
* Hyperglycemia
* Thyroid disease
* Metabolic disease
* Type I or Type II Diabetes
* Use of anabolic-androgenic steroids
* Use of antioxidant supplements, NSAIDS, or nutritional supplements known to stimulate recovery or muscle mass gains, heart disease, prescription medications, dietary supplements that enhance muscle strength or muscle recovery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2020-03-02 (Actual); Primary Completion 2020-06-12 (Actual); Study Completion 2020-06-12 (Actual)

PRIMARY OUTCOMES:
Changes in Blood Markers of Muscle Damage | Baseline, Week 5, Post-Week 5
  Experimental outcome examining blood protein concentrations in fasted whole blood samples.This outcome will be analyzed for the entire study population and will be analyzed as a sub-analysis in females only.
- Changes in subjective recovery scale that is directly related to recovery and inversely related to soreness. | Immediately prior to every resistance training session throughout the study.
  Assessed through a visual analog scale numbered 0-10 with visual descriptors. This outcome will be analyzed for the entire study population and will be analyzed as a sub-analysis in females only.

SECONDARY OUTCOMES:
Changes in Muscle Power | Baseline, Week 5, Post-Week 5
  Assessed through ground reaction forces during countermovement- and squat-jumps on a force plate. This outcome will be analyzed for the entire study population and will be analyzed as a sub-analysis in females only.
Changes in Muscle Strength | Baseline, Week 5, Post-Week 5
  Assessed by isometric mid-thigh pull. This outcome will be analyzed for the entire study population and will be analyzed as a sub-analysis in females only.
Changes in Salivary Immunoglobulin A | Baseline, Week 5, Post-Week 5
  Experimental outcome examining the concentration of IgA in fasted saliva samples. This outcome will be analyzed for the entire study population and will be analyzed as a sub-analysis in females only.
Changes in Body Composition | Baseline, Post-Week 5
  Body Composition will be assessed via dual-energy x-ray absorptiometry (DXA). Using this method, changes in total-, lean-, and fat-mass will be examined. This outcome will be analyzed for the entire study population and will be analyzed as a sub-analysis in females only.
Changes in Superoxide Dismutase (SOD) | Baseline, Week 5, Post-Week 5
  Experimental outcome examining superoxide dismutase in fasted whole blood samples. This is another protective antioxidant enzyme measured from whole blood. This outcome will be analyzed for the entire study population and will be analyzed as a sub-analysis in females only.

CONTACTS AND LOCATIONS:
Locations (1):
- The Applied Science and Performance Institute, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No
There are no intentions of sharing IPD with other researchers.